CLINICAL TRIAL: NCT00854217
Title: Cardioprotective Effects of Endogenous Erythropoietin in Patients Undergoing Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Mona Momeni, MD, Cliniques Universitaires saint Luc
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/03FEV/047
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- placebo, hemodilution (Placebo Comparator)
  Interventions: Procedure: acute normovolemic hemodilution

INTERVENTIONS:
Procedure: acute normovolemic hemodilution

SUMMARY:
Several studies have highlighted the cardioprotective effects of acute normovolemic hemodilution during cardiac surgery. The aim of our study is to show that an increase in endogenous erythropoietin (EPO) might explain the cardioprotective effects of acute normovolemic hemodilution against ischemia-reperfusion phenomena.

DETAILED DESCRIPTION:
The major physiologic function of EPO is thought to be the induction of erythropoiesis. However, a growing body of evidence indicates that EPO has tissue-protective effects and prevents tissue damage during ischemia. In an ex vivo proof-of-concept, protective effects of EPO have been shown in human myocardium.

Several studies have demonstrated that acute normovolemic hemodilution before aortic cross clamping decreases perioperative myocardial damage. We hypothesized that the onset of acute anemia increases the endogenous EPO concentration, which explains the cardioprotective effects of acute normovolemic hemodilution.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 80 years old undergoing CABG with or without cardiopulmonary bypass

Exclusion Criteria:

* emergencies
* redo operations
* combined surgery
* men with Hb< 120g/dL and women with Hb< 110g/ dL
* patients with preoperative creatinine> 2.2 mg/dL
* poor ventricular function (EF < 50%)
* subjects with a pulmonary disease, hepatic disease
* subjects with carotid stenosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Decrease in Troponin -I values | 4 h

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires saint Luc, Brussels, Belgium

REFERENCES:
- [Background] Licker M, Sierra J, Kalangos A, Panos A, Diaper J, Ellenberger C. Cardioprotective effects of acute normovolemic hemodilution in patients with severe aortic stenosis undergoing valve replacement. Transfusion. 2007 Feb;47(2):341-50. doi: 10.1111/j.1537-2995.2007.01111.x. PMID 17302782
- [Background] Licker M, Ellenberger C, Sierra J, Kalangos A, Diaper J, Morel D. Cardioprotective effects of acute normovolemic hemodilution in patients undergoing coronary artery bypass surgery. Chest. 2005 Aug;128(2):838-47. doi: 10.1378/chest.128.2.838. PMID 16100176